CLINICAL TRIAL: NCT01756495
Title: A Single Center Phase 1 Double Blind Study to Evaluate the Effect of Losmapimod on Cardiac Conduction as Compared to Placebo and Moxifloxacin in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Losmapimod on Cardiac Conduction as Compared to Placebo and Moxifloxacin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 116628
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Acute Coronary Syndrome
Keywords: QTc,; GW856553 .; P38,
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Losmapimod 7.5 mg (Experimental): Each subject will receive losmapimod 7.5 mg BID orally for 5 days, in one of the 4 study periods (per randomization sequence) separated by a minimum washout period of 5 days
  Interventions: Drug: Losmapimod
- Losmapimod 20 mg (Experimental): Each subject will receive losmapimod 20 mg QD orally for 5 days, in one of the 4 study periods (per randomization sequence) separated by a minimum washout period of 5 days
  Interventions: Drug: Losmapimod
- Moxifloxacin 400 mg (Active Comparator): Each subject will receive moxifloxacin 400 mg orally on Day 5, in one of the 4 study periods (per randomization sequence) separated by a minimum washout period of 5 days
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator): Each subject will receive losmapimod matched placebo and moxifloxacin placebo orally for 5 days, in one of the 4 study periods (per randomization sequence) separated by a minimum washout period of 5 days
  Interventions: Drug: Losmapimod matched Placebo; Drug: Moxifloxacin Placebo

INTERVENTIONS:
Drug: Losmapimod — Wet granulation formulation, Film coated white, 7 mm round, biconvex, plain faced Tablet of 7.5 mg or 10 mg unit dose strength. Taken orally 7.5 mg BID / 20 mg QD for 5 days in one of the 4 study periods
  Arms: Losmapimod 20 mg; Losmapimod 7.5 mg
Drug: Moxifloxacin — 17.2mm x 7.1 mm capsule shaped pink biconvex tablet of 400 mg unit dose strength. Taken orally 400 mg on Day 5 in one of the 4 study periods
  Arms: Moxifloxacin 400 mg
Drug: Losmapimod matched Placebo — Direct compression formulation (visually matched to GW856553), Film coated white, 7 mm round, biconvex, plain faced Tablet. Taken orally for 5 days in one of the 4 study periods
  Arms: Placebo
Drug: Moxifloxacin Placebo — 16 mm x 8 mm capsule shaped to white film coated tablet. Taken orally for 5 days in one of the 4 study periods
  Arms: Placebo

SUMMARY:
This will be a double-blind, 4-period, randomized, cross-over study conducted in healthy adult subjects. The purpose of this study is to characterize the effect of orally administered losmapimod on the electrocardiogram (ECG) parameters with a focus on cardiac repolarization as measured by the corrected QT interval (QTc) duration, compared with placebo and moxifloxacin. Moxifloxacin (Avelox) is a drug with a known potential to create a mild QTc interval prolongation; therefore, it will serve as a positive control to validate the ability of this study to detect a change in the QTc interval. All subjects will participate in 4 study periods separated by a minimum washout period of 5 days. Each subject will receive one of 4 regimens (A = Losmapimod 7.5 milligram [mg] Twice daily [BID] x 5 days, B = Losmapimod 20 mg Once daily [QD] x 5 days, C = moxifloxacin 400 mg on Day 5, D = Losmapimod matched placebo and moxifloxacin placebo x 5 days) in each of the 4 planned study periods in a randomized, cross-over fashion. Subjects will be assigned to one of four treatment sequences following a Williams design (ABDC, BCAD, CDBA, DACB). Follow-up visit will occur 10 to 14 days after end of Period 4

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac safety monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GlaxoSmithKline (GSK) Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent
* A female subject is eligible to participate if she is of

  1. Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] >40 MIU/mL and estradiol <40 pg/mL [<147 pmol/L] is confirmatory)
  2. Child-bearing potential and is abstinent or agrees to use one of the allowed contraception methods with a failure rate of <1% (Oral contraceptive, either combined or progestogen alone, Injectable progestogen, Implants of etonogestrel or levonorgestrel, Estrogenic vaginal ring, Percutaneous contraceptive patches, Intrauterine device [IUD] or intrauterine system [IUS], Male partner sterilization [vasectomy with documentation of azoospermia] prior to the female subject's entry into the study, and this male is the sole partner for that subject, Male condom combined with a female diaphragm, either with or without a vaginal spermicide [foam, gel, cream or suppository], Male condom combined with a vaginal spermicide [foam, gel, cream or suppository]) for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit
* Body weight >=50 kg and Body mass index (BMI) within the range 19 to 28 kg/m^2 (inclusive)
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)

Exclusion Criteria:

* Subjects with cardiac conduction abnormalities on the screening 12-lead ECG denoted by any of the following

  1. QTcB or QTcF >450 msec
  2. PR interval >200 msec or <=110 msec
  3. evidence of second- or third- degree atrioventricular block (AVB)
  4. clinically significant pathological Q-waves (defined as Q-wave >40 msec or depth greater than 0.4 to 0.5 mV)
  5. evidence of ventricular pre-excitation
  6. electrocardiographic evidence of complete left bundle branch block (LBBB), right bundle branch block (RBBB), incomplete LBBB
  7. intraventricular conduction delay with QRS duration >110 msec
  8. bradycardia as defined by sinus rate <45 beats per minute (BPM) or tachycardia as defined by sinus rate >100 BPM
* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination or ECG
* Subjects with a personal or family history of QTc prolongation, symptomatic cardiac arrhythmias or cardiac arrest
* History of hypersensitivity to moxifloxacin or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen
* A positive test for Human immunodeficiency virus (HIV) antibody result within 3 months of screening
* History of regular alcohol consumption within 6 months of the study defined as (For US sites) an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Pregnant females as determined by positive serum human chorionic gonadotropin (hCG) test at screening or prior to dosing
* Lactating females
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated
* History of sensitivity to heparin or heparin-induced thrombocytopenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01-10 (Actual); Primary Completion 2013-04-23 (Actual); Study Completion 2013-04-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QT interval corrected for heart rate by Fridericia's formula (QTcF) at each time point for losmapimod 20 mg QD on Day 5 as compared with time matched placebo | Baseline and Day 5 of the corresponding study period
  Triplicate ECGs will be collected at three baseline pre-dose time points (at -45 min, -30 min and -15 min) on Day 1 of the corresponding study period. Period baseline will be the average of triplicate pre-dose assessments. Triplicate Holter ECGs measurements will be evaluated at 14 post-dose time points (0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 and 24 hours) on Day 5 of the corresponding study period and will be averaged prior to calculation of changes from period baseline and statistical analyses

SECONDARY OUTCOMES:
Change from baseline in QTcF at each time point for losmapimod 7.5 mg BID on Day 5 as compared with time-matched placebo | Baseline and Day 5 of the corresponding study period
  Triplicate ECGs will be collected at three baseline pre-dose time points (at -45 min, -30 min and -15 min) on Day 1 of the corresponding study period. Period baseline will be the average of triplicate pre-dose assessments. Triplicate Holter ECGs measurements will be evaluated at 14 post-dose time points (0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 and 24 hours) on Day 5 of the corresponding study period and will be averaged prior to calculation of changes from period baseline and statistical analyses
Change from baseline in QTcF at each time point for moxifloxacin 400 mg single dose as compared with time-matched placebo | Baseline and Day 5 of the corresponding study period
  Triplicate ECGs will be collected at three baseline pre-dose time points (at -45 min, -30 min and -15 min) on Day 1 of the corresponding study period. Period baseline will be the average of triplicate pre-dose assessments. Triplicate Holter ECGs measurements will be evaluated at 14 post-dose time points (0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 and 24 hours) on Day 5 of the corresponding study period and will be averaged prior to calculation of changes from period baseline and statistical analyses
Change from baseline in QT interval corrected for heart rate by Bazett's formula (QTcB) at each time point for losmapimod (7.5 mg BID and 20 mg QD) and moxifloxacin (400 mg) on Day 5 as compared with time matched placebo | Baseline and Day 5 of all 4 study period
  Triplicate ECGs will be collected at three baseline pre-dose time points (at 45 min, -30 min and -15 min) on Day 1 of all study periods. Period Baseline will be the average of triplicate pre-dose assessments. Triplicate Holter ECGs measurements will be evaluated at 14 post-dose time points (0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 and 24 hours) on Day 5 of all the study period and will be averaged prior to calculation of changes from period baseline and statistical analyses
Change from baseline at each time point on Day 5 for other cardiac electrophysiological parameters: QT, PR, QRS, heart rate (HR) and ECG waveform morphology for losmapimod (7.5 mg BID and 20 mg QD) and moxifloxacin | Baseline and Day 5 of all 4 study period
  Single 12-lead ECG that automatically calculates the heart rate and measures PR, QRS, QT will be taken at 0, 2, 4 and 6 hour time points
Area under the plasma concentration-time curve (AUC) of losmapimod and its metabolite GSK198602 at doses of 7.5 mg BID and 20 mg QD, as well as 400 mg single dose of moxifloxacin | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 and approximately 24 hours post-dose on Day 5 of all 4 study period
  Pharmacokinetics (PK )Trough samples will be collected pre-dose on Days 3 and 4 of each period
Maximum observed plasma concentration (Cmax) of losmapimod and its metabolite GSK198602 at doses of 7.5 mg BID and 20 mg QD, as well as 400 mg single dose of moxifloxacin | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 and approximately 24 hours post-dose on Day 5 of all 4 study period
  PK Trough samples will be collected pre-dose on Days 3 and 4 of each period
Time to Cmax (Tmax) of losmapimod and its metabolite GSK198602 at doses of 7.5 mg BID and 20 mg QD, as well as 400 mg single dose of moxifloxacin | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18 and approximately 24 hours post-dose on Day 5 of all 4 study period
  PK Trough samples will be collected pre-dose on Days 3 and 4 of each period
Model parameters appropriate for concentration-QT analysis of losmapimod, metabolite and moxifloxacin (e.g. slope and intercept) | Day 5 of all 4 study period
  The relationship between losmapimod as well as GSK198602 plasma concentrations following repeat oral administration and the time-matched drug-placebo difference in QTc interval (∆∆QTc) will be explored graphically. If an apparent concentration-effect relationship exists, a population PK/ (pharmacodynamics) PD model will be established using nonlinear mixed effects modeling techniques with NONMEM software
Physical examination findings to assess safety and tolerability of losmapimod and moxifloxacin | Up to Day 49
  A complete physical examination (of the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen [liver and spleen], lymph nodes and extremities, height and weight) will occur at the screening and follow up visits. A brief physical examination (of the skin, lungs, cardiovascular system, and abdomen [liver and spleen]) will occur at Day -1
12-lead ECGs measurements to assess safety and tolerability of losmapimod and moxifloxacin | Up to Day 49
  As part of safety assessments, single 12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals
Clinical laboratory test measurements to assess safety and tolerability of losmapimod and moxifloxacin | Up to Day 49
  Samples will be collected at Screening, Day -1, follow-up for assessing safety
Clinical monitoring/observation | Up to Day 49
  The safety and tolerability of repeat oral doses of losmapimod 20mg QD and 7.5mg BID, as well as a single dose of moxifloxacin
Number of subjects with adverse events | Up to Day 49
  The safety and tolerability will be assessed by adverse events (AEs) of repeat oral doses of losmapimod 20mg QD and 7.5mg BID, as well as a single dose of moxifloxacin
Blood pressure measurements to assess safety and tolerability of losmapimod and moxifloxacin | Up to Day 49
  One measurement of blood pressure will be taken at Screening, Day -1 and Follow Up at the 0 hour timepoint on Day -1 and Follow up. Blood pressure measurement will be taken at 0, 2, 4 and 6 hour time points on Days 1, 4 and 5
HR measurements to assess safety and tolerability of losmapimod and moxifloxacin | Up to Day 49
  One measurement of HR will be taken at Screening, Day -1 and Follow Up at the 0 hour timepoint on Day -1 and Follow up. HR measurement will be taken at 0, 2, 4 and 6 hour time points on Days 1, 4 and 5

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116628 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116628?search=study&search_terms=116628#rs
- Available data/document: Study Protocol: 116628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register